CLINICAL TRIAL: NCT03897959
Title: FOLEY VERSUS KOHLI FOR SUPRAPUBIC CATHETER ASSOCIATED PROBLEMS STUDY
Brief Title: COMPARISON OF KOHLI AND FOLEY CATHETERS IN SUPRAPUBIC CATHETER PATIENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nellie Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KVF2019
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Catheter Infection; Complications; Catheter
Keywords: suprapubic, urinary catheter

STUDY DESIGN:
Intervention Model Description: Patients will utilize existing urinary drainage catheter for 30 days and then switch to alternative for 30 days. Patient will repeat this cycle once more.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Kohli vs Foley Study (Other): Compare various performance characteristics of two urinary catheters.
  Interventions: Device: Kohli vs Foley catheter

INTERVENTIONS:
Device: Kohli vs Foley catheter — Alternative suprapubic catheter used for bladder drainage.

SUMMARY:
The purpose of this medical research study is to compare two different urinary drainage catheters to see which has fewer problems with blockages and pain. The study involves completing 16 weekly 3-question surveys either online or by phone. The new catheters are FDA-approved and will be provided for FREE. No medications will be given.

DETAILED DESCRIPTION:
The purpose of this study is to see if a redesign of the catheter to remove the extended tip of the conventional urinary catheter will reduce problems with catheter blockage or catheter-associated discomfort. By eliminating the extended tip, the bladder wall will no longer be subject to the tip rubbing on the bladder wall. This could lead to fewer problems with blockages and less irritation and trauma to the bladder lining. A reduction in trauma to the bladder wall could reduce pain, bladder inflammation/irritation and the risk of urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Indwelling suprapubic Foley urinary catheter for at least 30 days prior to entry with anticipation for continued indwelling urinary catheterization for at least 30 days after entry into the study.
* Catheter associated discomfort or difficulty with mucous plugging of the catheter.

Exclusion Criteria:

* Inability to provide informed consent
* No catheter associated discomfort or problems with mucous plugging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Suprapubic catheter blockage - failure to drain | 1 year
  To determine whether an indwelling suprapubic low profile Kohli Atraumatic Catheter causes less patient-reported mucous plugging than a traditional indwelling suprapubic Foley catheter.

SECONDARY OUTCOMES:
Suprapubic catheter pain | 1 year
  To determine whether an indwelling suprapubic low profile Kohli Atraumatic Catheter causes less patient-defined discomfort than a traditional indwelling suprapubic Foley catheter. Pain will be accessed using a Visual Analog Pain scale.
Suprapubic catheter urinary tract infection (UTI) | 1 year
  To determine whether an indwelling suprapubic low profile Kohli Atraumatic Catheter reduces catheter-associated urinary tract infections (CAUTI's) than a traditional indwelling suprapubic Foley catheter. Patient symptoms such as hematuria, lower abdomen discomfort, frequent, painful urination, and pelvic pressure will be used to diagnose the presence of UTI.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Urogynecology, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No